CLINICAL TRIAL: NCT04987138
Title: Safety and Effectiveness Study of the Zenflow Spring System - A Minimally Invasive Treatment for LUTS Associated With BPH
Brief Title: Safety and Effectiveness Study of the Zenflow Spring System
Acronym: BREEZE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zenflow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-0130
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: BPH (Benign Prostatic Hyperplasia); Lower Urinary Tract Symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, multinational, 2:1 randomized, single-blinded, controlled clinical trial of the Zenflow Spring System. Following unblinding, control patients may elect to receive treatment with the Zenflow Spring System or exit the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient and site personnel administering follow-up assessments to 3 months will be blinded to the study assignment. Unblinding will occur at 3 months post procedure after follow-up assessments are completed.
  All patients will be asked post-treatment if they believe they are in the Treatment Arm, Control Arm, or do not know. The blinding questionnaire will be administered at discharge and at the 1-month and 3-month follow-up assessments.
  Control Arm patients can receive treatment with the Zenflow Spring System within 30 days after their 3-month follow-up assessments are completed, and their symptoms warrant treatment and enrollment criteria are met.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Roll-in Cohort (Other): Each Investigator will be allowed to treat up to 3 roll-in subjects with the Spring Implant prior to initiation of randomization. Roll-in patients will be followed for 60 months.
  Interventions: Device: Zenflow Spring System
- Treatment Arm (Active Comparator): Includes all patients who are randomized and start the treatment procedure. During the procedure the patient will be shielded from the treatment area and cystoscopy screen. The patient and site personnel administering follow-up assessments will be blinded to the study arm through the 3-month follow-up visit. Unblinding will occur at 3 months post-procedure after the assessments are completed. Follow up will continue for 60 months.
  Interventions: Device: Zenflow Spring System
- Control Arm (Sham Comparator): Includes all patients who receive a sham procedure. Patients will be shielded from the treatment area and cystoscopy screen. A Foley Catheter is placed into the patient's bladder and inflated. Additionally, devices will be used to produce mock deployment sounds of the Zenflow procedure. Once complete, the balloon will be deflated and the catheter will be removed, completing the procedure. Control arm subjects are followed for 3 months and exited from the study unless they elect and qualify for Crossover.
  Interventions: Device: Sham Procedure
- Crossover Cohort (Other): Control Arm (Sham) patients can receive treatment with the Zenflow Spring System after their 3-month follow-up assessments are completed, and their symptoms warrant treatment and enrollment criteria are met. The study visit follow-up schedule will restart and the subject will be followed for 60 months post Zenflow Spring implantation. Unless treated with the Spring System, the subject will be exited from the study once they have completed their 3-month follow-up visit.
  Interventions: Device: Zenflow Spring System

INTERVENTIONS:
Device: Zenflow Spring System — The Zenflow Spring Implant is an electropolished and passivated nickel titanium alloy (nitinol) implant. The implant is constructed from a single wire strand formed into ring elements connected by spine sections. There are four sizes of implants ranging from 16 mm to 24 mm in length and 14 mm to 16 mm in diameter to implant in the subject's prostatic urethra. The implant is placed in the urethra using a custom delivery catheter and cystoscope (Spring Scope). The implant is intended to be permanent but can be removed if necessary.
  Arms: Crossover Cohort; Roll-in Cohort; Treatment Arm
Device: Sham Procedure — A18 Fr Foley Catheter is placed into the patient's bladder. To mimic the Treatment Arm procedure, the Foley Catheter balloon will be inflated in the bladder. Once inflated, slight tension will be applied against the subject's bladder neck. While tension is being applied the site staff will follow a script to simulate the Zenflow procedural steps. Additionally, devices will be used to produce mock deployment sounds of the Zenflow procedure. Once complete, the balloon will be deflated and the catheter will be removed, completing the procedure.
  Other Names: Foley Catheter
  Arms: Control Arm

SUMMARY:
Evaluate the safety and effectiveness of the Zenflow Spring System in relieving LUTS associated with BPH.

DETAILED DESCRIPTION:
Prospective, multi-center, multinational, 2:1 randomized, single-blinded, controlled clinical trial of the Zenflow Spring System.

Patients randomized to the treatment group will undergo Zenflow Spring placement.

Patients randomized to the control group will undergo a Sham procedure. Patients and site personnel administering follow-up assessments will be blinded to the randomized treatment through completion of the 3-month follow-up visit. Once a patient has completed their 3-month follow-up assessments, they will be unblinded. Following unblinding, patients who received a Sham procedure may elect to receive treatment with the Zenflow Spring System or alternatively they may exit the study.

The duration of study participation is 60 months for patients who receive a Spring Implant and 3 months for subjects in the Control Arm.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to comply with all the assessments of the study,
2. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate and has signed the informed consent form,
3. ≥ 45 years of age,
4. Baseline IPSS score ≥ 13; ≥ 1 in the IPSS voiding to storage sub-score ratio (IPSS-V/S),
5. Prostate volume 25 - 80 cc by transrectal ultrasound (TRUS), measured within 120 days post study consent,
6. Prostatic urethral length between 25 and 45 mm, as measured by cystoscopic pull-back,
7. Failed, intolerant, or subject choice to not take a medication regimen for the treatment of LUTS.

Exclusion Criteria:

1. Obstructive intravesical median prostatic lobe as determined by ultrasound (i.e., more than 10 mm intravesical prostatic protrusion on sagittal mid-prostate plane via abdominal ultrasound),
2. High bladder neck with the absence of lateral lobe encroachment indicating a high likelihood of primary bladder neck obstruction as determined by the Investigator,
3. Urethral stricture, meatal stenosis, or bladder neck stricture - either current or recurrent,
4. Anatomical anomalies that will not accommodate the Implant, as determined by cystoscopy (e.g., prostatic urethral length to height geometry),
5. Requires indwelling catheter or intermittent catheterization to void,
6. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer (Subjects with a PSA level above 2.5 ng/mL, or age specific, or local reference ranges should have prostate cancer excluded to the Investigator's satisfaction),
7. One of the following baseline test results, taken from a single uroflowmetry reading:

   1. Urinary volume void ≤ 125mL (pre-bladder urinary volume of ≥ 150 mL required),
   2. Peak urinary flow rate (Qmax) of ≤ 5 ml/second or > 15 mL/second,
   3. Post- void residual volume (PVR) > 250 mL
8. History of other diseases causing voiding dysfunction including urinary retention (e.g., uncontrolled diabetes, diagnosis of neurogenic bladder, Parkinson's disease, multiple sclerosis, etc.),
9. Subjects with overactive bladder in the absence of benign prostatic obstruction,
10. Acute urinary tract infection (UTI) or finding of asymptomatic bacteriuria (Note: subject can be enrolled if the UTI is treated and followed with a negative urine test result), or subjects with history of recurrent UTIs (defined as > 3 UTIs in the past 12 months),
11. Concomitant bladder stones,
12. Previous pelvic irradiation or radical pelvic surgery,
13. Previous prostate surgery, including: enucleation, resection, vaporization, thermotherapy, ablation, stenting or prostatic urethral lift,
14. Chronic prostatitis, recurrent prostatitis, chronic pelvic pain syndrome (CPPS), or painful bladder syndrome within the past 12 months
15. Known allergy to nickel,
16. Life expectancy less than 60 months,
17. Use of concomitant medications (e.g., anticholinergics, antispasmodics or tricyclic antidepressants) affecting bladder function,
18. Inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure (Note: low dose aspirin therapy (81 mg) is permitted),
19. Taking 5-alpha-reductase inhibitors within 3 months of baseline evaluation,
20. Taking one of the following within 2 weeks of baseline evaluation:

    1. alpha-blockers,
    2. imipramine,
    3. anticholinergics,
    4. cholinergic gonadotropin releasing hormonal analogues,
    5. Phosphodiesterase-5 Enzyme Inhibitors (Tadalafil) in doses for BPH,
    6. Beta-3 adrenergic receptor agonist (Mirabegron),
21. Taking androgens, unless eugonadal state for at least 3 months or greater as documented by the Investigator,
22. Taking one of the following within 24 hours of pre-treatment (baseline) evaluation:

    1. phenylephrine, or,
    2. pseudoephedrine,
23. Future fertility concerns, or,
24. In the Investigator's opinion, the subject has a physical, psychological, or medical impairment that might prevent study completion or would confound study results (including subject questionnaires).

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety - The need for urinary catheterization | Greater than 7 days after procedure
  The rate of extended post-operative urinary catheterization (> 7 days from treatment) for inability to void among patients treated with the Zenflow Spring System.
Safety - Adverse Events | Procedure through 12 months
  The rate of device or procedure related serious adverse events in both the Treatment Arm and the Sham Arm.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) as compared to Sham | Procedure to 3 months
  The Treatment Arm will be considered superior to the Control Arm (Sham) when the mean 3-month improvement from baseline score for the IPSS symptom questionnaire demonstrates a minimum statistical margin of 25% compared to mean improvement from baseline for the Control Arm (Sham) alone.
Effectiveness- Symptoms Improvement | Procedure to 12 months
  The mean percent change in IPSS in the treatment arm is at least 30% improvement over the Patient's pre-treatment baseline score.

SECONDARY OUTCOMES:
Safety - Adverse Events | Procedure through 60 months
  Rate of device or procedure related adverse events at all time points.
Safety - Pain Assessment Questionnaire | Procedure through 3 months
  Comparison of pain at discharge to 2-week, 1- and, 3-month follow-up visits per Visual Analogue Scale (VAS) questionnaire. The VAS questionnaire asks the patient to indicate on a scale of 1 to 10 his level of pain where 1 is no pain and 10 is the worst pain.
Safety - Sexual Health Questionnaire 1 | 3 months post procedure through 24 months post procedure
  Change in sexual health characterized by the questionnaire Sexual Health Inventory for Men (SHIM).
Safety - Sexual Health Questionnaire 2 | 3 months post procedure through 24 months post procedure
  Change in sexual health characterized by questionnaire Male Sexual Health Questionnaire - Ejaculatory Domain (MSHQ-EjD)
Safety - Device Removal | Procedure through 60 months
  Assessment of adverse events outcomes related to a Spring Implant removal procedure.
Safety - Classification of Adverse Events | Procedure through 3 months
  Proportion of patients with adverse events classified as Clavien-Dindo Grade IIIb or higher or any event resulting in persistent disability
Effectiveness - long term symptom improvement 1 | Procedure through 12 months
  Percent of patients who experience at least a 30 percent improvement in IPSS from their baseline pre-treatment score
Effectiveness - long term symptom improvement 2 | Procedure through 60 months
  Mean percent change in IPSS in the treatment arm compared to baseline at all timepoints other than the primary endpoints.
Effectiveness - flow metrics | 1 month post procedure through 60 months
  Change from baseline in uroflowmetry measures of peak flow rate (Qmax)
Effectiveness - Re-intervention (device) | Procedure through 60 months
  Post-procedure incidence of secondary reintervention using an alternate surgical LUTS therapy.
Effectiveness - Re-intervention (drug) | Procedure through 60 months
  Post-procedure incidence of secondary reintervention using standard pharmacological agents for LUTS therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roehrborn, M.D, Principal Investigator — UT Southwestern, Dallas, TX
Locations (7):
- United States (7):
  - American Institute of Research, Los Angeles, California
  - Northshore University Health System, Glenview, Illinois
  - Sheldon Freedman, MD, LTD, Las Vegas, Nevada
  - Carolina Urologic Research Associates, Myrtle Beach, South Carolina
  - Midtown Urology Associates, Austin, Texas
  - Urology Austin, PLLC, Austin, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No